CLINICAL TRIAL: NCT02719093
Title: Role of FSHR Polymorphism p.N680S in the Therapy With FSH in Patients Who Underwent Varicocele Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: U.O. Chirurgia Andrologica (Other)
Collaborators: Androcenter, Napoli, Italy (Other)
Responsible Party: Principal Investigator, Maurizio Carrino, Medical Doctor, Director of U.O. Chirurgia Andrologica, U.O. Chirurgia Andrologica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIRURGIAANDROLOGICA-1
Record Dates: First submitted 2015-12-12; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Infertility, Male; Varicocele
Keywords: Infertility Male; Receptors FSH; Varicocele; FSH therapy
MeSH Terms: conditions — Infertility, Male; Varicocele | interventions — follitropin beta; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- recombinant FSH (Experimental): recombinant FSH 150UI daily
  Interventions: Drug: recombinant FSH

INTERVENTIONS:
Drug: recombinant FSH — Subcutaneous injection
  Other Names: Puregon; Gonal-F

SUMMARY:
Two common SNPs are located in linkage disequilibrium in exon 10 of FSHR. The 2039 A>G variant is regularly analyzed to characterize the exon 10 haplotype. In the last years, it has been showed an influence of FSHR 2039 A>G on FSH levels, testicular volume, sperm concentration and the total sperm count. A recent Cochrane review showed a beneficial effect on live birth and pregnancy of gonadotrophin treatment for men with idiopathic male factor subfertility. Which FSHR polymorphism can benefit from FSH treatment is clinically very important, in particular for what regards nonidiopathic patients. In many andrological units, patients underwent adiuvant therapy with purified or recombinant FSH after varicocelectomy. FSH treatment in patients after varicocelectomy could improve spermatogenesis, but there aren't multicentric trials that confirm its validity. Usually, in our hospital only patients with a morphologic aspect of hypospermatogenesis underwent therapy with purified or recombinant FSH, because this therapy is not much useful in patient with Partial Sertoli-cell-only syndrome or maturation arrest. The purpose of our study is to correlate "non responder" patients who underwent FSH adiuvant therapy after varicocele surgery with a p.N680S FSHR polymorphism. Moreover the investigators suppose that "non responder" patients can beneficiate from a high-dose therapy with FSH. This is a prospective intervention study in which are recruited males with OligoAstenoTeratozoospermic (OAT) and varicocele. The partecipants will undergo subinguinal microsurgical varicocelectomy (Marmar technique) and needle aspiration testicular cytology (Foresta technique).

DETAILED DESCRIPTION:
Two common SNPs (c.919 A>G, pT307A, rs 6165 and c.2039 A>G, p.N680S, rs6166) are located in linkage disequilibrium in exon 10 of FSHR. The 2039 A>G variant is regularly analyzed to characterize the exon 10 haplotype.

It is well known that follice-stimulating hormone (FSH) receptor (FSHR) polymorphism p.N680S mediates different responses to FSH in vitro, and this polymorphism is associated with the ovarian response in controlled ovarian hyperstimulation. In the last years, FSHR gene polymorphisms have been studied as potential risk factors for spermatogenetic failure. It is shown an influence of FSHR 2039 A>G on FSH levels and testicular volume. Trends of higher FSH and lower testicular volume were observed in G-allele carriers (Ala307/Ser680). Men homozygous for Thr307/Asn680 had a lower mean serum FSH concentration compared with men with other genotypes. In addition, sperm concentrations and the total sperm counts were higher and their testes volumes were larger. Another clinical study showed that the patients with heterozygous Thr/Ala + Asn/Ser combined genotype were 2.65 times more susceptible to infertility than the control group. It is also shown the higher sensitivity of the receptor in FSHR 2039 A>G AA homozygotes1-2. A recent Cochrane review showed a beneficial effect on live birth and pregnancy of gonadotrophin treatment for men with idiopathic male factor subfertility. These study suggest that the analysis of this gene represents a valid pharmacogenetic approach to the treatment of male infertility, confirming also the importance of strict criteria for the selection of patients to be treated with FSH. Which FSHR polymorphism can benefit from FSH treatment is clinically very important, in particular for what regards nonidiopathic patients. It is also relevant from a pharmacoeconomic point of view. In many andrological units, patients underwent adiuvant therapy with purified or recombinant FSH after varicocelectomy. FSH treatment in patients after varicocelectomy could improve spermatogenesis, but there aren't multicentric trials that confirm its validity. Usually, in our hospital only patients with a morphologic aspect of hypospermatogenesis underwent therapy with purified or recombinant FSH, because this therapy is not much useful in patient with Partial Sertoli-cell-only syndrome or maturation arrest. The purpose of our study is to correlate "non responder" patients who underwent FSH adiuvant therapy after varicocele surgery with a p.N680S FSHR polymorphism. Moreover the investigators suppose that "non responder" patients can beneficiate from a high-dose therapy with FSH.

This is a prospective intervention study in which are recruited males with OligoAstenoTeratozoospermic (OAT) and varicocele. The partecipants will undergo subinguinal microsurgical varicocelectomy (Marmar technique) and needle aspiration testicular cytology (Foresta technique). One-hundred patients with a morphologic aspect of hypospermatogenesis at testicular cytology will take recombinant follitropin alfa 150UI i.m. 3 times/week for at least three month. At 3th month the partecipants will have a semen analyses, without interrupting the treatment, and the FSHR gene polymorphism p.N680S characterization with PCR in high resolution melting HRM from DNA extracted by a simple blood sample. Patients who will have a significative increase in at least two parameters of semen, will be considered "responders" while patients in which semen parameters will not improve or worsen will be considered "non responders". "Responders" patients will interrupt their therapy and will have a new semen analyses at six month to verify the maintenance of their semen parameters after only three months of therapy. "Non responders" patients will take a daily dose of rFSH 150 UI for additional three months, because the investigators suppose that men with specific polymorphisms who don't response to therapy need an higher dose to stimulate spermatogenesis and to have a spontaneous pregnancy. At 6th month also these patients will have a new semen analyses in order to verify if there are some improvements in their spermatogenesis.

ELIGIBILITY:
Inclusion Criteria:

* OligoAstenoTeratozoospemic patient: Spermatozoa < 15 x 106/ml, Motility < 32%, <4% normal forms

Exclusion Criteria:

* Medications and psychoactive or anabolic drugs in last six months.
* Alcohol abuse in last three months.
* Systemic disease(liver cirrhosis, renal failure or others).
* Exposure to pelvic radiation, cytotoxic agent or exposure to environmental toxins.
* Testicular dysgenesis, cryptorchidism or genetic abnormalities (karyotype, Y-chromosome deletions)
* No trauma, testicular torsion, previous orchitis, previous testicular tumors, surgery that can compromise vascularisation of the testes and lead to testicular atrophy, cryptorchidism or genitourinary infection in last one year.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Total sperm count | After subinguinal microsurgical varicocelectomy and therapy with recombinant follitropin alfa 150UI i.m. 3 times/week for three months
  Response to therapy indicated by significant increase in sperm count (million/ejaculate) according to WHO Laboratory Manual for the Examination and Processing of Human Semen (5th edn.)
Sperm concentration | After subinguinal microsurgical varicocelectomy and therapy with recombinant follitropin alfa 150UI i.m. 3 times/week for three months
  Response to therapy indicated by significant increase in sperm concentration (million/mL) according to WHO Laboratory Manual for the Examination and Processing of Human Semen (5th edn.)
Total motility | After subinguinal microsurgical varicocelectomy and therapy with recombinant follitropin alfa 150UI i.m. 3 times/week for three months
  Response to therapy indicated by significant increase in total motility (%) according to WHO Laboratory Manual for the Examination and
Progressive motility | After subinguinal microsurgical varicocelectomy and therapy with recombinant follitropin alfa 150UI i.m. 3 times/week for three months
  Response to therapy indicated by significant increase in progressive motility (%) according to WHO Laboratory Manual for the Examination and
Sperm morphology (normal forms) | After subinguinal microsurgical varicocelectomy and therapy with recombinant follitropin alfa 150UI i.m. 3 times/week for three months
  Response to therapy indicated by significant increase in sperm morphology (normal forms) (%) according to WHO Laboratory Manual for the Examination and

SECONDARY OUTCOMES:
Total sperm count | After a daily dose of rFSH 150 UI for additional three months in "non responders" patients to the first three months of therapy with recombinant follitropin alfa 150UI i.m. 3 times/week
  Response to therapy indicated by significant increase in sperm count (million/ejaculate) according to WHO Laboratory Manual for the Examination and
Sperm concentration | After a daily dose of rFSH 150 UI for additional three months in "non responders" patients to the first three months of therapy with recombinant follitropin alfa 150UI i.m. 3 times/week
  Response to therapy indicated by significant increase in sperm concentration (million/mL) according to WHO Laboratory Manual for the Examination and
Total motility | After a daily dose of rFSH 150 UI for additional three months in "non responders" patients to the first three months of therapy with recombinant follitropin alfa 150UI i.m. 3 times/week
  Response to therapy indicated by significant increase in total motility (%) according to WHO Laboratory Manual for the Examination and
Progressive motility | After a daily dose of rFSH 150 UI for additional three months in "non responders" patients to the first three months of therapy with recombinant follitropin alfa 150UI i.m. 3 times/week
  Response to therapy indicated by significant increase in progressive motility (%) according to WHO Laboratory Manual for the Examination and
Sperm morphology (normal forms) | After a daily dose of rFSH 150 UI for additional three months in "non responders" patients to the first three months of therapy with recombinant follitropin alfa 150UI i.m. 3 times/week
  Response to therapy indicated by significant increase in sperm morphology (normal forms) (%) according to WHO Laboratory Manual for the Examination and

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Carrino, Study Director — AORN A.CARDARELLI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tuttelmann F, Laan M, Grigorova M, Punab M, Sober S, Gromoll J. Combined effects of the variants FSHB -211G>T and FSHR 2039A>G on male reproductive parameters. J Clin Endocrinol Metab. 2012 Oct;97(10):3639-47. doi: 10.1210/jc.2012-1761. Epub 2012 Jul 12. PMID 22791757
- [Result] Casarini L, Moriondo V, Marino M, Adversi F, Capodanno F, Grisolia C, La Marca A, La Sala GB, Simoni M. FSHR polymorphism p.N680S mediates different responses to FSH in vitro. Mol Cell Endocrinol. 2014 Aug 5;393(1-2):83-91. doi: 10.1016/j.mce.2014.06.013. Epub 2014 Jun 23. PMID 24970684